CLINICAL TRIAL: NCT06629831
Title: The Effect of Preoperative Laboratory Values on Prognostic Factors Following Cytoreductive Surgery for Ovarian Cancer: Neutrophil to Lymphocyte Ratio, Platelet to Lymphocyte Ratio, Lymphocyte to Monocyte Ratio
Brief Title: Systemic Inflammatory Biomarkers in Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Duygu Akyol, Principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: 2024-59
Record Dates: First submitted 2024-09-27; First posted 2024-10-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Ovarian Cancer
Keywords: systemic inflammatory markers; ovarian cancer; cytoreductive surgery
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Population Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing cytoreduction surgery for ovarian cancer: Patients undergoing cytoreduction surgery for ovarian cancer
  Interventions: Other: group with complications; Other: group without complications

INTERVENTIONS:
Other: group with complications — Complications in patients undergoing cytoreduction surgery for ovarian cancer
Other: group without complications — Complications in patients undergoing cytoreduction surgery for ovarian cancer

SUMMARY:
In cancer patients, prognostic markers are needed to improve the management and clinical course of both the cancer itself and surgery therefor. Elevated systemic inflammatory markers are associated with morbidity and mortality in most cancer types. In this study, the investigators aimed to determine the prognostic value of inflammatory markers such as neutrophil to lymphocyte ratio (NLR), platelet to lymphocyte ratio (PLR), and lymphocyte to monocyte ratio (LMR) in patients undergoing cytoreductive surgery for ovarian cancer.

DETAILED DESCRIPTION:
Major gynaecological cancer surgery is a procedure with high complication rates and mortality risk due to both the patient' s old age and comorbidities and the extent of the surgery. Among such surgeries, ovarian cancer-related surgery has the highest mortality rate. Despite advances in early drug therapy and improvements in the cytotoxicity of drugs, ovarian cancer is frequently diagnosed at advanced stages, which further increases morbidity and mortality rates. Although many years have passed, the prognostic role of cytoreductive surgery on survival in ovarian cancers continues to be important. Predicting postoperative outcomes in these surgeries may reduce the length of hospital stay, need for stay in the intensive care unit, complications, and mortality. Therefore, the role of systemic inflammatory biomarkers needs to be comprehensively investigated to understand the carcinogenic mechanisms better.

For this purpose, the investigators planned to evaluate the prognostic effect of systemic inflammatory biomarkers on postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age

Exclusion Criteria:

* Patients with acute or inflammatory diseases
* Patients with hematological malignancies
* Patients with autoimmune diseases patients who underwent intraoperative hyperchemotherapy (HIPEC)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: A total of 187 patients who were operated in the gynecologic surgical oncology clinic in one year were retrospectively evaluated.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
the rate of systemic inflammatory biomarkers | up to 24 hours postoperative
  the investigator planned to evaluate the prognostic effect of systemic inflammatory biomarkers on postoperative complications.

CONTACTS AND LOCATIONS:
Locations (1):
- BasaksehiCam and Sakura City Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He W, Yin C, Guo G, Jiang C, Wang F, Qiu H, Chen X, Rong R, Zhang B, Xia L. Initial neutrophil lymphocyte ratio is superior to platelet lymphocyte ratio as an adverse prognostic and predictive factor in metastatic colorectal cancer. Med Oncol. 2013 Mar;30(1):439. doi: 10.1007/s12032-012-0439-x. Epub 2013 Jan 10. PMID 23307251
- [Background] Oreskov KO, Jensen KK, Gogenur I, Godthaab C, Jorgensen AB, Oreskov JO, Burcharth J, Ekeloef S. Limited value of preoperative neutrophil-to-lymphocyte ratio to predict post-operative outcomes after major emergency abdominal surgery. Dan Med J. 2021 Aug 20;68(9):A09200689. PMID 34477095
- [Background] Forget P, Dinant V, De Kock M. Is the Neutrophil-to-Lymphocyte Ratio more correlated than C-reactive protein with postoperative complications after major abdominal surgery? PeerJ. 2015 Jan 13;3:e713. doi: 10.7717/peerj.713. eCollection 2015. PMID 25653901
- [Background] Lapchak PH, Kannan L, Ioannou A, Rani P, Karian P, Dalle Lucca JJ, Tsokos GC. Platelets orchestrate remote tissue damage after mesenteric ischemia-reperfusion. Am J Physiol Gastrointest Liver Physiol. 2012 Apr 15;302(8):G888-97. doi: 10.1152/ajpgi.00499.2011. Epub 2012 Feb 2. PMID 22301111